CLINICAL TRIAL: NCT03302715
Title: KOLBIBAKT; The Association Between the Microbiological Environment in Colon and Colorectal Disease
Brief Title: The Association Between the Microbiological Environment in Colon and Colorectal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ulf Oskar Gustafsson, MD, PhD, Consultant Surgeon, associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KOLBIBAKT; 2017;1
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Microbial Colonization and Colorectal Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Consecutive cohort study with mucosal samples during colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mucosal biopsies (Experimental): Only blood samples and mucosal biopsies
  Interventions: Genetic: Mucosal tissue sampling

INTERVENTIONS:
Genetic: Mucosal tissue sampling — Mucosal tissue sampling for DNA analysis

SUMMARY:
Colorectal illness contributes significantly to the global burden of disease. Cancer, inflammatory bowel disease and diverticulosis result in substantial patients suffering and health care expenditures. The causes of colorectal diseases remain unclear.

New data suggests that intestinal bacteria may play a major role in the causal chain for many diseases, and the research on the microbial environment in the colon in relation to bowel disease is increasingly intense although the possibility for analysis of the composition of bacteria in the gut has so far been limited. However, new analytic methods based on powerful DNA sequencing, opens new opportunities.

In the surgical clinic at Danderyds hospital, Stockholm, 2500 colonoscopies are performed per year. The investigators have created a biobank with mucosal samples from patient's large bowel and will consecutively include all patients scheduled for colonoscopy during one year (N=2500). Biopsies from the colonic mucosa will be analysed in collaboration with the Clinical Genomics, Science for Life laboratory (Karolinska Institutet).

In Phase 1, the association between specific bacteria and colorectal disease will be investigated (hypothesis generating phase). In Phase 2, the investigators aim to identify specific bacterial biomarkers that could be used as screening tools, and lay the ground for future new treatments for colorectal disease.

Early detection and new treatment regimes would result in both significant patient benefits as well as reductions in healthcare costs.

DETAILED DESCRIPTION:
Project description Overall hypothesis: The colonic microbial environment correlates with bowel pathology and is relevant to development and progress of colorectal disease.

Research questions and outcomes:

In Phase 1 (year 1, hypothesis generating phase), the association between specific bacteria and the following diseases will be investigated: colorectal disease (colorectal cancer /polyps, adenomas (pre-cancerous lesions), inflammatory bowel disease (IBD) and diverticulosis).

Research questions:

1. Is the microenvironment of the gut mucosa in and around tissue with adenomas/colorectal adenocarcinoma, IBD and diverticulosis colonized with a bacterial set different from healthy mucosa?
2. Does age, sex and life/dietary habits impact different types of bacterial composition?

In Phase 2 (year 2-3), we aim to identify specific bacterial biomarkers that could be used as screening tools, and lay the ground for future new treatments for colorectal disease.

Primary research questions:

1. Are specific bacterial sets associated with early formation of adenoma and colorectal cancer?
2. Can these bacteria be used as faecal biomarkers in a colorectal screening program for cancer or be identified by serological biomarkers?
3. Can the identification of specific bacteria lead to further studies on the possible genesis of the emergence and growth of colorectal cancer?

Secondary research questions:

1. Are specific bacterial sets associated with IBD and diverticulosis and can those be used as faecal or serological biomarkers for disease?
2. Can treatment of these bacteria or their metabolites reduce the incidence of morbidity in relation to IBD or diverticulitis (inflammation in diverticula)?

Study population and implementation

Phase 1: (2017) -2018. During one year, all patients scheduled for colonoscopy at Danderyd's Hospital (sample size = 2500 patients) will be consecutively invited to participate in the study and to give informed consent.

Exclusion criteria: Bleeding risk (defined as a International Normalized Ratio (INR) > 1.6), severe dementia or inability to understand information and make an informed decision about participation.

Patients who agree to participate will receive an information letter about the study by mail (2-3 weeks before colonoscopy). In addition all patients will also receive a phone call as a reminder of the study. Before bowel preparation, patients will be asked to leave a faeces sample that will be saved for culture. Study participants will also be asked to complete a validated questionnaire on medical history, previous illnesses, diet, lifestyle habits, previous colonoscopies and antibiotic treatment. Immediately before the colonoscopy examination, four blood samples will be taken: Two for the analysis of HbA1c, haemoglobin and C-reactive protein (CRP) and two for storage at hospital's biobank robot for later analysis of biomarkers.

During colonoscopy, tissue samples in addition to routine diagnostic tissue samples will be taken from the colonic mucosa:

1. Two biopsies (one for DNA sequencing, one for cultivation) will be taken from a healthy part of colonic mucosa (preferably in the first part of the colon) in all patients.
2. Four biopsies, two (DNA + culture) from pathologic colonic mucosa (polyp (adenomas) / colorectal cancer / IBD/diverticulosis) and two (DNA + culture) in the nearby area of the pathologic mucosa.

Phase 2: 2018-2020.

1. Detection and investigation of biologically important bacteria and their metabolites (metagenomics and metabolomics (studies of chemical processes involving metabolites)) will be carried out for information about specific bacterial genes.
2. This data will then be statistically analysed for any association with various colorectal conditions, adjusting for confounding and exposures available in medical records and in the patient questionnaire (See below). These analyses will provide us with important novel information about the pathogenic mechanisms of relevance for development of cancer and inflammation.
3. Based on these expected findings of specific bacterial compositions in relation to colonic disease, specific disease mechanisms can begin to be analysed.
4. The possibilities of using disease-specific bacterial compositions as a clinical marker of colonic disease will also be explored. During this sub-study we will look at the association between mucosal microbiota and the microbiota in the feces. Thus, stool samples from all patients will be will be used to explore whether these correspond to the bacterial composition of the colonic mucosa sampled from the pathologic and healthy intestinal area. In addition, serological biomarkers will be examined in relation to specific bacterial compositions in mucosal samples from pathologic mucosa in all study patients.

Samples and analysis The samples are first stored and recorded in the Danderyd Hospital biobank and will thereafter be sent for DNA analysis at the Science for Life laboratory, Karolinska Institutet. The DNA analysis (primary variables) relates to massive parallel sequencing of the 16S rRNA gene that gives information about the composition of bacteria in the sample and the relative amount of bacteria down to the gene level. The results are presented as a diversity index (Shannon diversity index or alpha diversity within the same sample) and Unifrac analysis based on the software QIIME. The latter analysis shows differences in bacterial composition between samples - so-called beta diversity. In addition to16S sequencing, so called metagenomic sequencing will be performed on selected samples - with this assay one can also get information about the specific bacterial gene content and thus gain knowledge of pathogenic mechanisms with relevance to include cancer development. The validated questionnaire of diet and lifestyle habits will be analysed in relation to the microbial environment (dependent variable in this laboratory analysis).

ELIGIBILITY:
Inclusion Criteria:

* All colonoscopy cases

Exclusion Criteria:

* Not able to understand Swedish or to understand patientinformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Bacterial diversity in colorectal disease | 3 years
  DNA sequencing on mucosal sampling

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, Professor, Study Chair — Department of Surgery, Ersta Hospital, & Department of Clinical Sciences, Danderyd Hospital, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Not decided
Supporting Information: Study Protocol